CLINICAL TRIAL: NCT04520035
Title: A Prospective, Single Arm, Single Center, Phase II Clinical Trial of Neoadjuvant Chemotherapy With Camrelizumab in Locally Advanced Esophageal Squamous Cell
Brief Title: Neoadjuvant Chemotherapy With Camrelizumab in Locally Advanced Esophageal Squamous Cell
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jialei Wang, Principal Investigator, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMRE-CHEM-01
Record Dates: First submitted 2020-08-12; First posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: PFS
MeSH Terms: interventions — camrelizumab; Paclitaxel; Cisplatin; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neoadjuvant chemotherapy with camrelizumab (Experimental): paclitaxel and cisplatin
  Carilizumab 200 mg, every 3 weeks, 2 cycles.
  Paclitaxel 175 mg / m2, D1, every 3 weeks, 2 cycles
  Cisplatin 75mg / m2 D1, conventional hydration for 3 days, every 3 weeks, 2 cycles
  Interventions: Drug: camrelizumab; Drug: Paclitaxel; Drug: Neoadjuvant Chemotherapy

INTERVENTIONS:
Drug: camrelizumab — Carilizumab 200 mg, every 3 weeks, 2 cycles.Paclitaxel 175 mg / m2, D1, every 3 weeks, 2 cycles
  Other Names: Paclitaxel; Cisplatin
Drug: Paclitaxel — Cisplatin 75mg / m2 D1, conventional hydration for 3 days, every 3 weeks, 2 cycles
Drug: Neoadjuvant Chemotherapy — Neoadjuvant Chemotherapy

SUMMARY:
A prospective, single arm, single center, phase II clinical trial of neoadjuvant chemotherapy with camrelizumab in locally advanced esophageal squamous cell,to evaluate the progression free survival

ELIGIBILITY:
Inclusion Criteria:

1. The age ranged from 18 to 75 years 2. Middle or lower thoracic esophageal carcinoma 3. Gastroscopy showed squamous cell carcinoma 4. The clinical stage was c-txn1-3m0 5. ECOG score was 0-1 6. Can eat semifluid 7. Weight loss less than 20% in 6 months 8. Sign the consent form before treatment 9. One week before enrollment, the organ function level reached the following standards:

1. Bone marrow function: hemoglobin ≥ 100g / L, WBC ≥ 4.0 * 10 ^ 9 / L, neutrophil count ≥ 1.8 * 10 ^ 9 / L, platelet count ≥ 100 * 10 ^ 9 / L;
2. Liver: serum total bilirubin level ≤ 1.5 times normal upper limit value, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 1.5 times normal upper limit value;
3. Kidney: serum creatinine level is lower than 1.5 times of normal upper limit value or creatinine clearance rate ≥ 60ml / min, urea nitrogen ≤ 200mg / L;
4. Blood glucose: within the normal range and / or patients with diabetes are under treatment, but the blood glucose is controlled in a stable state;
5. Lung function: baseline FEV1 should be at least 2L; if the baseline FEV1 < 2L, it should be evaluated by surgical experts, and FEV1 > 800ml after surgery should be predicted;
6. Cardiac function: no myocardial infarction within 1 year; no unstable angina pectoris; no symptomatic severe arrhythmia; no cardiac insufficiency.

Exclusion Criteria:

1. The pathological findings were complex squamous cell carcinoma, including squamous adenocarcinoma, squamous cell carcinoma, carcinosarcoma, sarcomatoid carcinoma, etc
2. He had a history of subtotal gastrectomy
3. Patients with secondary primary cancer at the same time
4. The patients with distant metastasis indicated by imaging before treatment
5. Except for skin basal cell carcinoma, skin squamous cell carcinoma and / or cervical carcinoma in situ after effective treatment
6. Patients who have received chemoradiotherapy in the past
7. There were signs of esophageal perforation
8. Pregnant women of childbearing age
9. The patient has any active autoimmune disease or history of autoimmune disease (such as interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, etc.)
10. There are patients with the following active infectious diseases, including active pulmonary tuberculosis, active hepatitis B (HBV DNA ≥ 500 IU / ml), hepatitis C (hepatitis C antibody positive, and HCV-RNA higher than the detection limit of the analysis method), and known human immunodeficiency virus (HIV) infection
11. Those who are known to have bleeding diseases or other uncontrollable diseases and are unable to receive surgical treatment
12. Findings of physical examination or clinical trials that the researchers believe may interfere with the results or increase the risk of treatment complications for patients
13. Function of each organ of the patient:Previous interstitial lung disease, drug-induced interstitial disease, radiation pneumonitis requiring hormone therapy, or any active interstitial lung disease with clinical evidence, CT scan at baseline found the presence of idiopathic pulmonary fibrosis; uncontrolled massive pleural effusion or pericardial effusion;
14. Unstable systemic concomitant diseases (active infection, moderate to severe chronic obstructive pulmonary disease, poorly controlled hypertension, unstable angina pectoris, congestive heart failure, myocardial infarction within 6 months, severe mental disorders requiring drug control, liver, kidney or other metabolic diseases, neuropsychiatric diseases such as Alzheimer's disease);
15. Poor gastrointestinal function, absorption syndrome and active peptic ulcer;
16. Have received any of the following treatments:

1) Have received anti-PD-1 or anti-PD-L1 antibody treatment in the past; 2) Received any research drug within 4 weeks before the first use of the study drug; 3) At the same time, they were enrolled in another clinical study, unless it was an observational (non intervention) clinical study or an intervention clinical study follow-up; 4) Have received any anti-tumor treatment related to esophageal cancer, including but not limited to radiotherapy, chemotherapy, surgery, ESD, EMR, immunotherapy, targeted therapy, and traditional Chinese medicine treatment; 5) Subjects who needed systemic treatment with corticosteroids (10 mg prednisone equivalent dose per day) or other immunosuppressants within 2 weeks before the first use of the study drug were excluded from the use of corticosteroids for local esophageal inflammation and prevention of allergy, nausea and vomiting. Other special circumstances, need to communicate with the sponsor. In the absence of active autoimmune disease, inhaled or topical corticosteroids and corticosteroids with dose > 10 mg / day prednisone were allowed to be used instead; 6) Those who have received anti-tumor vaccine or received live vaccine within 4 weeks before the first administration of the study drug; 7) Major surgery or severe trauma occurred within 4 weeks before the first use of the study drug; 17. History of congenital or acquired immunodeficiency disease or organ transplantation; 18. He had a history of allergy to monoclonal antibodies, paclitaxel, cisplatin and other platinum drugs;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (pCR) | from the first cycle of treatment (day one) to two month after the last cycle (each cycle is 21 days)
  Pathological complete response rate

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer hospital Fudan University, Shanghai, Xuhui, China